CLINICAL TRIAL: NCT02243618
Title: The Effect of Proton Pump Inhibitor and Polaprezinc Combination Therapy for Healing of Endoscopic Submucosal Dissection-induced Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0381
Record Dates: First submitted 2014-09-15; First posted 2014-09-18 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2016-12

CONDITIONS: Gastric Adenoma; Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — polaprezinc; rebamipide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebamipide group (Active Comparator)
  Interventions: Drug: Rebamipide
- Polaprezinc group (Active Comparator)
  Interventions: Drug: Polaprezinc

INTERVENTIONS:
Drug: Polaprezinc — Administration of pantoprazole 40 mg q.d. and polaprezinc 75 mg b.i.d. for 4 weeks after the ESD.
  Arms: Polaprezinc group
Drug: Rebamipide — Administration of pantoprazole 40 mg q.d. and rebamipide 100 mg t.i.d. for 4 weeks after the ESD.
  Arms: Rebamipide group

SUMMARY:
Endoscopic submucosal dissection (ESD) is an advanced technique that enables en bloc resection of superficial tumors in the gastrointestinal tract. ESD, however, is a time-consuming procedure that requires a high level of endoscopic skill to achieve a desirable oncologic outcome. Several procedure-related complications may occur after ESD. Especially, iatrogenic ulcer bleeding after ESD can be a concern for both endoscopists and patients. In order to reduce the bleeding rate, proton pump inhibitors (PPIs) are administered after ESD. In addition, ulcer protective agents such as rebamipide can be added to PPIs for accelerating ulcer healing. We aimed to evaluate the efficacy of polaprezinc for healing of iatrogenic ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 19 and 79
2. Patients with gastric adenoma or early gastric cancer
3. Patients with ECOG-PS 0 or 1
4. Patients with adequate renal function
5. Patients with adequate hepatic function
6. Patients with adequate bone marrow function

Exclusion Criteria:

1. Patients who has taken the medications for ulcer including PPIs, H2 blockers, and mucosal protective agents within 3 months prior to the ESD.
2. Patients who has taken steroid or NSAIDswithin 3 months prior to the ESD.
3. Patients who has undergone gastrostomy
4. Patients with allergy for pantoprazole, polaprezinc, or rebamipide.
5. Pregnant or breast feeding.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-14 (Actual)

PRIMARY OUTCOMES:
Ulcering healing rate | 4 weeks after the ESD
  Healing rate of the iatrogenic ulcer according to the type of ulcer protective agents (polaprezinc vs. rebamipide).

SECONDARY OUTCOMES:
Scarring change rate | 4 weeks after the ESD
  Scarring change rate of the iatrogenic ulcer according to the type of ulcer protective agents (polaprezinc vs. rebamipide).

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hospital, Seoul, South Korea